CLINICAL TRIAL: NCT00246142
Title: A 16-week Prospective Randomised Double-blind Study on Facilitation of DYSPORT® Effect on Myofascial Pain Syndrome (MPS) by Electrical Stimulation.
Brief Title: A Study of the Combination of Electrical Stimulation and Dysport® in Myofascial Pain Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-38-52120-104
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Myofascial Pain Syndromes
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to determine whether electrical stimulation enhances the effect of botulinum toxin type A (Dysport®) on myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck and shoulder pain for at least 6 months, refractory with other conservative treatments
* Presents at baseline with pain score greater than 50mm on 100mm length VAS. Pain score will be measured as overall pain over the 7 days preceding the visit during activities
* Active trigger point (TrP) defined as a tender spot localised in a taut band of muscle fibres associated with tenderness AND referred pain recognised by the patient into well-defined areas that are remote from the TrP area at palpation AND preferably local twitch response at palpation AND/OR jump sign at palpation

Exclusion Criteria:

* Disc/bone disease
* History of surgery on neck
* Neurological deficits, neuromuscular junction disorder, Motor Neuron disease
* Patient has received anesthetic injections to the target trigger point within 4 weeks of study enrolment, or corticosteroid injections within 3 months
* Systemic inflammatory disease
* Hypersensitivity to Dysport®
* Diffuse tender points, or diagnosed with fibromyalgia
* Previous electrical stimulation
* Previous injection of Dysport® within 6 months of study enrolment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06-27 (Actual); Study Completion 2007-06-27 (Actual)

PRIMARY OUTCOMES:
Changes in mean pain measured by Visual Analogue Scale (VAS) will be assessed. | Comparison of VAS will be performed before Dysport® injection and at 16 weeks after injection
Number of patients in percentage whose pain intensity measured by VAS decreases to less than 50% of baseline. | Before Dysport® injection and at 16 weeks after injection

SECONDARY OUTCOMES:
Pain threshold measured by pressure algometer. | At each visit
Neck Pain and Disability scale (NPAD) and Global Assessment of Impairment Scale (GAS) will be assessed. | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo HG, Bang MS, Chung SG, Jung SH, Lee SU. Effect of electrical stimulation on botulinum toxin a therapy in patients with chronic myofascial pain syndrome: a 16-week randomized double-blinded study. Arch Phys Med Rehabil. 2013 Mar;94(3):412-8. doi: 10.1016/j.apmr.2012.09.034. Epub 2012 Nov 1. PMID 23123438